CLINICAL TRIAL: NCT06734676
Title: Study of Multi-Modal Imaging Technology in MRI-Guided Transcranial Magnetic Stimulation Treatment for Parkinson's Disease
Brief Title: fMRI-guided Transcranial Magnetic Stimulation Treatment for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changping Laboratory (Other)
Collaborators: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PDHNTMS
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2023-05

CONDITIONS: Parkinson's Disease
Keywords: TMS; Parkinson's disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCAN (Experimental): 14-day iTBS on personalized SCAN localized by precision functional mapping
  Interventions: Device: Intermittent theta burst stimulation (iTBS)
- Effector (Active Comparator): 14-day iTBS on personalized effector-specific network localized by precision functional mapping
  Interventions: Device: Intermittent theta burst stimulation (iTBS)

INTERVENTIONS:
Device: Intermittent theta burst stimulation (iTBS) — iTBS: 90% RMT, 50Hz intraburst frequency, 3 pulses per burst, 5Hz interburst frequency, 2 seconds on/8 seconds off, totaling 1800 pulses over approximately 10 minutes. Each day includes 4 iTBS sessions (1800 pulses per session) with 50-minute intervals, totaling 7200 pulses per day for 14 consecutive days (100800 pulses total).

SUMMARY:
The goal of this clinical trial is to compare the efficacy of targeting the newly discovered SCAN versus traditional effector-specific networks in M1 using multimodal imaging and rTMS in patients with Parkinson's disease. The main question it aims to answer is: Is rTMS targeting the SCAN more effective than rTMS targeting effector networks?

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder commonly affecting middle-aged and elderly individuals. Besides conventional treatments such as medication (e.g., levodopa) and surgery (e.g., deep brain stimulation), non-invasive neuromodulation techniques, such as transcranial magnetic stimulation (TMS), have been widely used as a safe and well-tolerated non-pharmacological adjunct therapy for PD patients. However, the limited efficacy of TMS may be attributed to an incomplete understanding of PD-related cortical circuits and imprecise targeting.

Historically, the primary motor cortex (M1) has been selected as the repetitive TMS (rTMS) target for PD treatment. In 2022, Gordon et al. discovered a new network within the M1 that differs from effector-specific networks responsible for executing movements of specific body parts, such as those for the foot, hand, and face. This newly identified network, named the somato-cognitive action network (SCAN), is located in inter-effector regions and is responsible for motor planning, control, and coordination. Damage to this network correlates with key PD symptoms, making SCAN a promising new target for PD intervention.

This study aims to compare the efficacy of targeting the newly discovered SCAN versus traditional effector-specific networks in M1 using multimodal imaging and Intermittent theta burst stimulation (iTBS), a rapid form of rTMS. The objective is to provide new clinical evidence for non-invasive neuromodulation in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary PD per the MDS Clinical Diagnostic Criteria (2015) or the Chinese Parkinson's Disease Diagnostic Criteria (2016).
* Age 18-75.
* Stable use of anti-PD medication for at least two months prior to enrollment.
* Normal cognitive function (MMSE > 24).
* Understanding of the study and signing of informed consent.

Exclusion Criteria:

* Diagnosed with other neurological diseases, such as stroke, brain tumor, traumatic brain injury, motor neuron disease, Alzheimer's disease, multiple sclerosis, etc.
* Implanted medical devices incompatible with MRI, such as deep brain stimulators, pacemakers, cochlear implants, or vagus nerve stimulators.
* Conditions contraindicated for MRI, such as claustrophobia, tattoos, or magnetic metal implants.
* Personal or family history of epilepsy.
* Prior neuromodulation treatments (e.g., TMS, transcranial electrical stimulation, transcranial ultrasound stimulation) within the last three months.
* Other health abnormalities that the investigator deems unsuitable for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
MDS-UPDRS-III | Baseline, 7 days, 14 days
  The primary outcome is the difference in MDS-UPDRS-III scores at the "on" state at day 7 and day 14 after iTBS intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, PhD, Study Chair — Changping Laboratory
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data will be available to researchers upon reasonable request by contacting the corresponding authors after the publication of relevant papers.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: after the publication of relevant papers
Access Criteria: researchers upon reasonable request by contacting the corresponding authors

REFERENCES:
- [Background] Gordon EM, Chauvin RJ, Van AN, Rajesh A, Nielsen A, Newbold DJ, Lynch CJ, Seider NA, Krimmel SR, Scheidter KM, Monk J, Miller RL, Metoki A, Montez DF, Zheng A, Elbau I, Madison T, Nishino T, Myers MJ, Kaplan S, Badke D'Andrea C, Demeter DV, Feigelis M, Ramirez JSB, Xu T, Barch DM, Smyser CD, Rogers CE, Zimmermann J, Botteron KN, Pruett JR, Willie JT, Brunner P, Shimony JS, Kay BP, Marek S, Norris SA, Gratton C, Sylvester CM, Power JD, Liston C, Greene DJ, Roland JL, Petersen SE, Raichle ME, Laumann TO, Fair DA, Dosenbach NUF. A somato-cognitive action network alternates with effector regions in motor cortex. Nature. 2023 May;617(7960):351-359. doi: 10.1038/s41586-023-05964-2. Epub 2023 Apr 19. PMID 37076628
- [Background] Latorre A, Rocchi L, Berardelli A, Bhatia KP, Rothwell JC. The use of transcranial magnetic stimulation as a treatment for movement disorders: A critical review. Mov Disord. 2019 Jun;34(6):769-782. doi: 10.1002/mds.27705. Epub 2019 Apr 29. PMID 31034682
- [Background] Zhang W, Deng B, Xie F, Zhou H, Guo JF, Jiang H, Sim A, Tang B, Wang Q. Efficacy of repetitive transcranial magnetic stimulation in Parkinson's disease: A systematic review and meta-analysis of randomised controlled trials. EClinicalMedicine. 2022 Jul 29;52:101589. doi: 10.1016/j.eclinm.2022.101589. eCollection 2022 Oct. PMID 35923424